CLINICAL TRIAL: NCT06609278
Title: Culturally AdapTed Harm Reduction Intervention: Community Engaged InterVention for Black Adults That MisusE Opioids and Stimulants
Brief Title: THRIVE: Culturally AdapTed Harm Reduction Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brittany Miller-Roenigk (Other)
Collaborators: University of Cincinnati (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Brittany Miller-Roenigk, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 96815; UL1TR001998 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use; Stimulant Use
Keywords: Harm Reduction; Opioid Overdose; Stimulant Misuse; Opioid Misuse; Narcan; Fentanyl Test Strips
MeSH Terms: conditions — Harm Reduction; Opiate Overdose; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THRIVE (Experimental): Participants will complete pre- and post-intervention quantitative measures assessing their motivation and comfort using Narcan and FTS. In addition, participants will also participate in a semi-structured qualitative focus group after completing the intervention session to assess harm reduction needs in their community, additional barriers participants expect with the adapted intervention, feasibility of the intervention, and perceived knowledge of opioid overdose and prevention and intervention tools gained from prior to the intervention to afterwards.
  Interventions: Behavioral: harm reduction intervention

INTERVENTIONS:
Behavioral: harm reduction intervention — Each participant will complete a pre-test at Study Visit 1 prior to the intervention, participate in the intervention, then complete a post-test. After the intervention, participants will participate in a recorded focus group. Participants will be offered FTS, Narcan, first aid supplies at the study visit.

SUMMARY:
The goal of this study is to develop and test a culturally adapted harm reduction intervention among Black adults who misuse opioids and/or stimulants. The questions it aims to answer include: will the culturally adapted harm reduction educational intervention increase overall knowledge of overdose and prevention/intervention techniques and increase confidence and willingness to use/teach interventions to others at-risk.

DETAILED DESCRIPTION:
The overall study design is a mixed methods pilot developing and testing a culturally adapted intervention to enhance knowledge about and motivation to use opioid overdose harm reduction strategies, including Fentanyl Test Strips (FTS) and Narcan. Given the preliminary nature of this pilot study designed to develop an adapted intervention, subjects will not be randomized and there will be no control group or placebo.

Aim 1 is a qualitative design in which investigators will conduct two focus group sessions with a group of up to 8 Black adults who have misused opioids and stimulants in the past 30 days. Participants will be recruited to have about 50% gender and age representation across four cohorts: born 1996-2006; born 1985-1995; born 1974-1984; and born 1960-1973; with one male and one female in each cohort. A semi-structured qualitative focus group format will be utilized for each focus group session to allow for flexibility in asking additional questions based on participant responses. Individuals are excluded if they do not want to be audio-recorded, since a main component of the study is recording focus groups. Aim 1 will occur in Louisville, KY and full study visits will be recorded.

Aim 2 is a cross-sectional mixed method design in which the culturally adapted intervention developed during Aim 1 will be piloted after institutional review board (IRB) modification approval of the intervention among about 48-60 Black adults residing in Louisville, KY and Cincinnati, OH. Each study site will recruit three groups of up to 8-10 participants to pilot the intervention, resulting in approximately 6 groups and 48-60 participants. Eligible participants for Aim 2 are aged 18-65 and will be recruited to have approximately 50% male and female members overall but not specific to age cohorts. Participants will complete pre-and post-intervention quantitative measures assessing their motivation and comfort using Narcan and Fentanyl Test Strips (FTS). In addition, participants will also participate in a semi-structured qualitative focus group after completing the intervention session to assess harm reduction needs in their community, additional barriers participants expect with the adapted intervention, feasibility of the intervention, and perceived knowledge of opioid overdose and prevention and intervention tools gained from prior to the intervention to afterwards. Individuals are excluded if they do not want to be audio-recorded, since a main component of the study is recording focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black or African American
* Currently a resident of study areas
* Report misuse of stimulants and/or opioids in the last six months

Exclusion Criteria:

* Do not identify as Black or African American
* If they participated in Aim 1 of the study
* Do not want to be audio-recorded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Change in participant confidence using harm reduction techniques | Baseline and post intervention (approximately 2 hours)
  Confidence will be measured by a pre - post test survey with a Likert type scale measured from 1 (not confident) to 10 (very confident).
Change in participant willingness to use harm reduction techniques | Baseline and post intervention (approximately 2 hours)
  Willingness will be measured by a pre - post test survey with a Likert type scale measured from 1 (not willing) to 10 (very willing).
Change in participant comfort to possess harm reduction techniques | Baseline and post intervention (approximately 2 hours)
  Comfort will be measured by a pre - post test survey with a Likert type scale measured from 1 (not comfortable) to 10 (very comfortable).
Change in participant confidence describing how to use harm reduction techniques to others | Baseline and post intervention (approximately 2 hours)
  Confidence will be measured by a pre - post test survey with a Likert type scale measured from 1 (not confident) to 10 (very confident).
Change in participant willingness to teach others how to use harm reduction techniques | Baseline and post intervention (approximately 2 hours)
  Willingness will be measured by a pre - post test survey with a Likert type scale measured from 1 (not willing) to 10 (very willing).

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Miller-Roenigk, PhD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Louisville Central Community Center, Louisville, Kentucky
  - Urban Minority Alcoholism and Drug Abuse Outreach Program (UMADAOP) of Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT06609278/ICF_000.pdf